CLINICAL TRIAL: NCT03641339
Title: Defining Skin Immunity of a Bite of Key Insect Vectors in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 180139; 18-I-0139
Record Dates: First submitted 2018-08-21; First posted 2018-08-22 (Actual); Results first posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2019-08

CONDITIONS: Zika; Dengue; Malaria; Chikungunya; Leishmaniasis
Keywords: Mosquito; Saliva; Immune Response; Sand Fly; Biopsy
MeSH Terms: conditions — Zika Virus Infection; Dengue; Malaria; Chikungunya Fever; Leishmaniasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A: One vector feeding and three biopsies (Experimental): Undergo one vector feeding and three biopsies on Day 0
  Interventions: Other: One vector feeding
- Cohort B: Four vector feedings and three biopsies (Experimental): Undergo 4 vector feedings over 8 weeks and 3 biopsy procedures after the 4th and final feeding
  Interventions: Other: Four vector feeding

INTERVENTIONS:
Other: One vector feeding — Participants will undergo one feeding by one of three colony- reared vectors (Aedes aegypti mosquitos, Anopheles gambiae mosquitos, or Lutzomyia longipalpis sand flies)
  Arms: Cohort A: One vector feeding and three biopsies
Other: Four vector feeding — Participants will undergo four feedings by one of three colony- reared vectors (Aedes aegypti mosquitos, Anopheles gambiae mosquitos, or Lutzomyia longipalpis sand flies), each about 2 weeks apart, with the same vector type.
  Arms: Cohort B: Four vector feedings and three biopsies

SUMMARY:
Background:

Mosquitoes and similar insects called sand flies carry parasites that can cause diseases. These viruses and parasites can spread quickly and be difficult to control. How people s bodies respond to insect bites may affect how they get infected. The response to bites is caused by the immune system, which helps fight off infections. Researchers want to study the immune response in skin to mosquito or sand fly bites and how the response changes after bites on multiple days. This may help researchers develop better vaccines.

Objective:

To study the immune response in skin to certain insect bites and how that changes after bites on multiple days.

Eligibility:

Healthy adults ages 18-64

Design:

Participants will be screened under another protocol. Women must agree to practice effective contraception or abstinence. All participants must agree to not donate blood or use certain lotions or creams on visit days.

Some participants will have 2 visits over a week. Others will have 5 visits over 8 weeks.

All participants will have the following at least once:

Medical history

Physical exam

Blood and urine collected

Mosquito or sand fly feeding. Up to 10 insects will feed on participant s arm for up to 20 minutes. The insects are grown at NIH and do not carry any diseases. The skin will be checked and bites will be treated.

Skin samples taken. The skin will be cleaned and numbed. A tool will remove a small piece of skin from 3 places on the arm.

About a week after the last visit, participants will be called to see how they feel.

DETAILED DESCRIPTION:
Vector-borne diseases continue to cause significant morbidity and mortality worldwide despite ongoing control efforts. Vectors like sand flies and mosquitoes deliver the pathogen into the skin of humans while taking a blood meal. Most vaccines under development ignore the importance of the complex infectious inoculum delivered by the vector and the local immune response that occurs at the site of the bite. In addition, many preclinical studies are carried out in animal models that do not replicate the natural route of infection, transmission by vector bites, and often bypass the skin interface altogether. As such, these studies do not evaluate what role the vector plays in the initiation of these infections. Further compounding this problem, many clinical studies are performed in naïve individuals who have never been exposed to the vector, while those living in endemic areas will have had long-term exposure to vectors through uninfected bites.

A cumulative body of evidence from animal models demonstrates that a variety of vector-derived components are co-delivered with the pathogen and may play an important role in the establishment of infection. There is limited knowledge of the effect of these vector-derived factors on the immune response in human skin and their potential impact on infection establishment.

In this protocol, we will examine the early skin immune response to bites of three arthropods: the mosquito Aedes aegypti, the vector of Zika, dengue, and chikungunya viruses; the mosquito Anopheles gambiae, the vector of malaria; and the sand fly Lutzomyia longipalpis, the vector of leishmaniasis. We will also explore how multiple vector bite exposures over time modulate future immune response at the bite site. Healthy participants will come to the National Institutes of Health (NIH) and undergo feeding by one of the three vectors, then have three skin punch biopsies performed by trained medical practitioners to evaluate local immune response. Participants in Cohort A will have one feeding; participants in Cohort B will have 4 feedings, each 2 weeks apart. Biopsies will be collected after the final feeding. Blood will be collected after the one feeding in Cohort A and after the fourth and final feeding in Cohort B to assess systemic immune response.

With the current rise of vector-borne diseases in the United States and around the world, we hope the results of this study contribute to future vaccine design and clinical development strategies for vector-borne diseases.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals must meet all of the following criteria to be eligible for study participation:

* Healthy women and men who are greater than or equal to 18 and less than or equal to 64 years of age.
* Able to provide informed consent.
* Willingness to complete all study visits and comply with all study requirements.
* Willing to have samples stored for future research.
* A female is eligible for this study if she meets 1 of the following:

  * Of non-childbearing potential (i.e., women who have had a hysterectomy or tubal ligation or are postmenopausal, as defined by no menses in greater than or equal to 1 year).
  * Of childbearing potential but agrees to practice effective contraception or abstinence for 4 weeks prior to enrollment through the completion of the study. Acceptable methods of contraception include a male partner who is sterile and is the sole sexual partner of the female participant or a male partner who uses a condom with spermicide plus 1 or more of the following that is used by the female: 1) implants of levonorgestrel; 2) injectable progestogen; 3) an intrauterine device with a documented failure rate of <1%; 4) oral contraceptives; and 5) double barrier method including diaphragm.
* Agrees to not use scented lotions, deodorants, or topical creams on each feeding day.
* Agrees to not take aspirin or any other NSAID within 7 days of a biopsy.
* Agrees to not use topical steroid creams or ointments throughout the study without prior permission of Principal Investigator (PI).
* Vector-specific antibody enzyme-linked immunosorbent assay (ELISA) to one of the three vectors (the one to which the individual is assigned) is <2.5 standard deviations above the negative control for Cohort A only.

EXCLUSION CRITERIA:

Individuals meeting any of the following criteria will be excluded from study participation:

* Any underlying or current medical condition that, in the opinion of the investigator, would interfere with participation in the study.
* Any participant that is HIV positive.
* A clinically significant (as determined by the PI) baseline Grade 1 or greater toxicity by the toxicity table.
* History of severe allergic reaction (including to mosquito or other insect bites) with generalized urticaria, angioedema, anaphylaxis, or anaphylactoid reaction.
* Prone to allergic responses and/or significant history of allergies, including seasonal or specific allergies as determined by the PI.
* Receipt of any investigational drug that is unlicensed within 3 months or 5.5 half- lives (whichever is greater) prior to enrollment.
* Receipt of any unlicensed vaccine within 6 months prior to enrollment.
* Self-reported or known history of alcoholism or drug abuse within 6 months prior to enrollment, or positive urine test for drugs of abuse at screening (excluding positive test for tetrahydrocannabinol (THC) or its metabolites if usage is less than 3 times per week).
* Self-reported or known history of psychiatric or psychological issues that require treatment and are deemed by the PI to be a contraindication to protocol participation.
* Any use of medications that affect blood clotting within 3 months, history of abnormal blood clotting, or result outside of the normal laboratory range for measurements of prothrombin time (PT), partial thromboplastin time (PTT), or international normalized ratio (INR) that may suggest a problem with blood clotting.
* History of significant scarring after previous biopsies, lacerations, abrasions, surgeries, or other skin procedures (e.g., cosmetic piercings) that are deemed by the PI to be a contraindication to protocol participation.
* Pregnant or breastfeeding.

Co-enrollment Guidelines: Co-enrollment in other trials is restricted, but may take place after consultation with the study staff and approval from the PI.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Memoli, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Fauci AS, Morens DM. Zika Virus in the Americas--Yet Another Arbovirus Threat. N Engl J Med. 2016 Feb 18;374(7):601-4. doi: 10.1056/NEJMp1600297. Epub 2016 Jan 13. No abstract available. PMID 26761185
- [Background] Edqvist PH, Fagerberg L, Hallstrom BM, Danielsson A, Edlund K, Uhlen M, Ponten F. Expression of human skin-specific genes defined by transcriptomics and antibody-based profiling. J Histochem Cytochem. 2015 Feb;63(2):129-41. doi: 10.1369/0022155414562646. Epub 2014 Nov 19. PMID 25411189
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-I-0139.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Exposure Cohort A: Aedes Aegypti: One vector feeding: Participants will undergo one feeding by Aedes aegypti mosquitoes and then three biopsies on Day 0 were performed
- Multiple Exposure Cohort B: Aedes Aegypti: Four vector feeding: Participants will undergo four feedings by Aedes aegypti mosquitos each about 2 weeks apart, with the same vector type. 3 biopsy procedures were performed after the 4th and final feeding
- Single Exposure Cohort A: Anopheles Gambiae: One vector feeding: Participants will undergo one feeding by Anopheles gambiae mosquitoes and then three biopsies on Day 0 were performed
- Multiple Exposure Cohort B: Anopheles Gambiae: Four vector feeding: Participants will undergo four feedings by Anopheles gambiae mosquitoes each about 2 weeks apart, with the same vector type. 3 biopsy procedures were performed after the 4th and final feeding
- Single Exposure Cohort A: Lutzomyia Longipalpis: One vector feeding: Participants will undergo one feeding by Lutzomyia longipalpis and then three biopsies on Day 0 were performed
- Multiple Exposure Cohort B: Lutzomyia Longipalpis: Four vector feeding: Participants will undergo four feedings by Lutzomyia longipalpis each about 2 weeks apart, with the same vector type. 3 biopsy procedures were performed after the 4th and final feeding
Period: Overall Study
Arm/Group | Single Exposure Cohort A: Aedes Aegypti | Multiple Exposure Cohort B: Aedes Aegypti | Single Exposure Cohort A: Anopheles Gambiae | Multiple Exposure Cohort B: Anopheles Gambiae | Single Exposure Cohort A: Lutzomyia Longipalpis | Multiple Exposure Cohort B: Lutzomyia Longipalpis
Started | 16 | 17 | 15 | 16 | 15 | 16
Completed | 15 | 15 | 15 | 14 | 15 | 15
Not Completed | 1 | 2 | 0 | 2 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who completed all study visits and sample collection.
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Exposure Cohort A: Aedes Aegypti | Multiple Exposure Cohort B: Aedes Aegypti | Single Exposure Cohort A: Anopheles Gambiae | Multiple Exposure Cohort B: Anopheles Gambiae | Single Exposure Cohort A: Lutzomyia Longipalpis | Multiple Exposure Cohort B: Lutzomyia Longipalpis | Total
Number analyzed (Participants) | 15 | 15 | 15 | 14 | 15 | 15 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.27 (8.36) | 30.67 (9.40) | 35.60 (9.66) | 33.07 (9.42) | 32.47 (11.62) | 32.73 (11.44) | 32.62 (9.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 12 | 9 | 8 | 11 | 11 | 57
  Male | 9 | 3 | 6 | 6 | 4 | 4 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 2 | 2 | 3 | 4 | 15
  Not Hispanic or Latino | 12 | 14 | 12 | 12 | 11 | 11 | 72
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 1 | 1 | 1 | 1 | 1 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 1 | 3 | 4 | 4 | 19
  White | 8 | 7 | 10 | 8 | 7 | 9 | 49
  More than one race | 2 | 2 | 3 | 1 | 1 | 0 | 9
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 2 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 15 | 14 | 15 | 15 | 89

OUTCOME MEASURES:

1. Primary Outcome: Number of Differentially Expressed Genes Between Bitten (Case) Versus Unbitten (Control) Skin for Each of the Three Vector Groups
Description: Number of differentially expressed genes between bitten and unbitten skin with adjusted p-values (adjusted for multiple comparisons) of < 0.05 and a minimum absolute fold change > 4 in samples derived from skin biopsies for the three vector groups - Aedes aegypti, Anopheles gambiae, Lutzomyia longipalpis
Time Frame: Up to 48 hours post bite
Population: Every participant who had skin biopsies.
Measure: Number; unit: number of differentially expressed genes
Arm/Group | Single Exposure Cohort A: Aedes Aegypti | Multiple Exposure Cohort B: Aedes Aegypti | Single Exposure Cohort A: Anopheles Gambiae | Multiple Exposure Cohort B: Anopheles Gambiae | Single Exposure Cohort A: Lutzomyia Longipalpis | Multiple Exposure Cohort B: Lutzomyia Longipalpis
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7 | 7
number of differentially expressed genes
  30 minutes post bite | 18 | NA — Participants in Cohort B did not have a 30 minute time point per study protocol | 1 | NA — Participants in Cohort B did not have a 30 minute time point per study protocol | 5 | NA — Participants in Cohort B did not have a 30 minute time point per study protocol
  4 hours post bite | 227 | 179 | 12 | 72 | 172 | 204
  48 hours post bite | NA — Participants in Cohort A did not have a 48 hour time point per study protocol. | 503 | NA — Participants in Cohort A did not have a 48 hour time point per study protocol | 982 | NA — Participants in Cohort A did not have a 48 hour time point per study protocol | 797

2. Primary Outcome: Participants With Local Skin Adaptive Immune Response After Multiple Exposures Over Time to Bites of Each of the Three Vector Groups
Description: Number of participants with certain types of inflammatory cell infiltrates, which includes neutrophils, mononuclear cells, and eosinophils, in the skin biopsies of bitten skin at 30 minutes, 4 hours, and 48 hours post bite for each of the three vector groups - Aedes aegypti, Anopheles gambiae, and Lutzomyia longipalpis
Time Frame: Up to 48 hours post bite
Population: Every participant who had skin biopsies.
Measure: Number; unit: participants
Arm/Group | Single Exposure Cohort A: Aedes Aegypti | Multiple Exposure Cohort B: Aedes Aegypti | Single Exposure Cohort A: Anopheles Gambiae | Multiple Exposure Cohort B: Anopheles Gambiae | Single Exposure Cohort A: Lutzomyia Longipalpis | Multiple Exposure Cohort B: Lutzomyia Longipalpis
Number analyzed (Participants) | 8 | 8 | 8 | 7 | 8 | 8
participants
  Neutrophils 30 minutes post bite | 3 | NA — Participants in Cohort B did not have a 30 minute time point per study protocol | 2 | NA — Participants in Cohort B did not have a 30 minute time point per study protocol | 0 | NA — Participants in Cohort B did not have a 30 minute time point per study protocol
  Mononuclear Cells 30 minutes post bite | 3 | NA — Participants in Cohort B did not have a 30 minute time point per study protocol | 1 | NA — Participants in Cohort B did not have a 30 minute time point per study protocol | 3 | NA — Participants in Cohort B did not have a 30 minute time point per study protocol
  Eosinophils 30 minutes post bite | 4 | NA — Participants in Cohort B did not have a 30 minute time point per study protocol | 0 | NA — Participants in Cohort B did not have a 30 minute time point per study protocol | 0 | NA — Participants in Cohort B did not have a 30 minute time point per study protocol
  Neutrophils 4 hours post bite | 5 | 6 | 1 | 3 | 3 | 3
  Mononuclear Cells 4 hours post bite | 5 | 3 | 0 | 2 | 2 | 6
  Eosinophils 4 hours post bite | 3 | 5 | 0 | 2 | 1 | 4
  Neutrophils 48 hours post bite | NA — Participants in Cohort A did not have a 48 hour time point per study protocol | 1 | NA — Participants in Cohort A did not have a 48 hour time point per study protocol | 0 | NA — Participants in Cohort A did not have a 48 hour time point per study protocol | 0
  Mononuclear Cells 48 hours post bite | NA — Participants in Cohort A did not have a 48 hour time point per study protocol | 8 | NA — Participants in Cohort A did not have a 48 hour time point per study protocol | 7 | NA — Participants in Cohort A did not have a 48 hour time point per study protocol | 8
  Eosinophils 48 hours post bite | NA — Participants in Cohort A did not have a 48 hour time point per study protocol | 4 | NA — Participants in Cohort A did not have a 48 hour time point per study protocol | 1 | NA — Participants in Cohort A did not have a 48 hour time point per study protocol | 2

ADVERSE EVENTS:
Time Frame: Monitoring for adverse events was over a 7 day period for all Cohort A groups. Monitoring for adverse events was over a 51 day period for all Cohort B groups.
Arm/Group | Single Exposure Cohort A: Aedes Aegypti | Multiple Exposure Cohort B: Aedes Aegypti | Single Exposure Cohort A: Anopheles Gambiae | Multiple Exposure Cohort B: Anopheles Gambiae | Single Exposure Cohort A: Lutzomyia Longipalpis | Multiple Exposure Cohort B: Lutzomyia Longipalpis
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/14 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/14 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 5/15 | 3/15 | 6/14 | 1/15 | 6/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Exposure Cohort A: Aedes Aegypti (N=15) | Multiple Exposure Cohort B: Aedes Aegypti (N=15) | Single Exposure Cohort A: Anopheles Gambiae (N=15) | Multiple Exposure Cohort B: Anopheles Gambiae (N=14) | Single Exposure Cohort A: Lutzomyia Longipalpis (N=15) | Multiple Exposure Cohort B: Lutzomyia Longipalpis (N=15)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drainage at biopsy site (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systolic hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feverish (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Latent Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coryza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URI (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema at biopsy site (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fractured metatarsal (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Difficulty sleeping (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
dry cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT03641339/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT03641339/ICF_001.pdf